CLINICAL TRIAL: NCT01490762
Title: A Phase 1, Open-label, Randomized, Crossover Design Clinical Trial in Healthy Normal Volunteers to Evaluate Insulin Exposure and Effect Following Inhalation of Technosphere® Insulin Inhalation Powder at Multiple Doses Using the Gen2C Inhaler
Brief Title: Healthy Normal Volunteers Looking at Exposure and Effects of Multiple Doses of Technosphere® Insulin (TI) Using the Gen2C Inhaler
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MKC-TI-176
Record Dates: First submitted 2011-12-05; First posted 2011-12-13 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Healthy
Keywords: PK; PD
MeSH Terms: interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regular Human Insulin (Active Comparator): Subcutaneous injection
  Interventions: Drug: Regular Human Insulin
- TI and Regular Human Insulin (Experimental): All subjects have 4 clamp procedures with 10, 30, 60,80 units of TI and 1 clamp with 15 IU Regular Human Insulin
  Interventions: Drug: Technosphere Insulin Inhalation Powder using the Gen2C inhaler

INTERVENTIONS:
Drug: Technosphere Insulin Inhalation Powder using the Gen2C inhaler — Inhalation Powder
  Arms: TI and Regular Human Insulin
Drug: Regular Human Insulin — Subcutaneous injection
  Arms: Regular Human Insulin

SUMMARY:
This is an open-Label, Randomized Study in Healthy Normal Volunteers looking at exposure and effects (PK/PD) of multiple doses of Technosphere® Insulin (TI) using the Gen2C inhaler.

DETAILED DESCRIPTION:
Healthy Normal Volunteers will be randomized to a sequence of 4 different doses of Technosphere® Insulin (TI), inhaled using the Gen2C device, and one dose of subcutaneously injected Regular Human Insulin. A euglycemic clamp procedure will be performed at each dosing visit. The purpose of this study is to determine the insulin dose proportionality/linearity of Technosphere® Insulin (TI) Inhalation Powder based on the AUCo-180 after administration of the following doses using the Gen2C inhaler:

* 10 U (one 10 U cartridge)
* 30 U (one 10 U and one 20 U cartridge)
* 60 U (three 20 U cartridges)
* 80 U (four 20 U cartridges)

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 55 years who are considered healthy based on screening physical examination, medical history, clinical chemistry, and urinalysis
* Good venous access for blood draws
* No smoking in the previous 6 months (including cigarettes, cigars, pipes) and negative urine cotinine testing (< 100 ng/mL)
* Body mass index (BMI) < 32 kg/m2
* FEV1 = 80% of the Third National Health and Nutrition Examination Survey (NHANES III) predicted
* FVC = 80% of the Third National Health and Nutrition Examination Survey (NHANES III) predicted
* Written informed consent provided

Exclusion Criteria:

* Blood donation of 500 mL within the previous 56 days
* Fasting blood sugar >130 mg/dL
* History of coronary artery disease, peripheral vascular disease, or congestive heart failure
* Allergy to study drug, food, or other study material (eg, peanuts, soy products)
* Clinically significant active or chronic illness
* History of asthma, COPD, or any other clinically relevant chronic lung disease
* Respiratory tract infection within 4 weeks before screening
* Donation of blood within 3 months before screening
* History of drug or alcohol abuse
* Positive urine drug screen
* Clinically significant screening ECG, physical examination, laboratory test, or vital sign abnormality
* Any subject who, in the opinion of the PI or a designee, appears to not be qualified for this study
* Exposure to any other investigational drug or device within 30 days before treatment or within 90 days before treatment for drugs known to modify glucose metabolism (except metformin
* History of malignancy within the 5 years before screening (other than basal cell carcinoma)
* History of human immunodeficiency virus (HIV) infection or hepatitis B or C
* Women who are pregnant, lactating, or planning to become pregnant during the clinical study period
* Any subject who at Visit 2 has a blood glucose value = 150 mg/dL 2 hours after the meal, should be discussed with the MKC medical monitor and may be removed as potentially having impaired glucose tolerance
* Inability, in the opinion of the PI or a designee, to adequately inhale TI Inhalation Powder
* Women of childbearing potential (defined as premenopausal and not surgically sterilized or postmenopausal for fewer than 2 years) not practicing adequate birth control. Adequate birth control is defined as using oral, percutaneous, or transdermal contraceptives; condoms and diaphragms (double barrier) with a spermicide; or intrauterine devices. Postmenopausal for the purposes of this clinical study includes experiencing amenorrhea for 2 or more years or being surgically sterile

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2011-12; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
area-under-the-serum insulin concentration versus time curve (AUC0-240min) for inhaled Technosphere Insulin (TI) post-dosing of a TI dose (10 U, 30 U, 60 U or 80U). Time points: 0, 5, 10, 15, 20, 30, 45, 60, 90, 120, 180 and 240 minutes post-TI dosing | crossover 4 times over the course of up to 5 weeks

SECONDARY OUTCOMES:
Area-under-the-serum insulin concentration versus time curve (AUC0-240min) for inhaled Technosphere Insulin (TI) compared to that of subcutaneous regular human insulin (RHI) | crossover 5 times over the course of up to 6 weeks
  Timepoints: 0, 5, 10, 15, 20, 30, 45, 60, 90, 120, 180 and 240 minutes after administration of TI dosing; 0, 15, 30, 60, 90, 120, 180, 240, 300, 360, 480 and 600 minutes after RHI dosing
Area-under-the-serum glucose infusion rate (GIR AUC0-240min) for TI compared to AUC0-600min for RHI | crossover 5 times over the course of up to 6 weeks
  Timepoints for TI: 0, 5, 10, 15, 20, 30, 45, 60, 90, 120, 180 and 240 minutes after TI dosing Timepoints: 0, 15, 30, 60, 90, 120, 180, 240, 300, 360, 480 and 600 minutes after RHI dosing
Safety variables included adverse events (AEs), clinical laboratory tests, vital signs and physical examinations | crossover 5 times for up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Chair — Mannkind Corporation
Locations (1):
- Profil Institute for Clinical Research, Chula Vista, California, United States